CLINICAL TRIAL: NCT05252091
Title: An Exploratory Clinical Study of Herombopag Olamine Tablets for Thrombocytopenia Induced by Chemotherapy Combined With Immunotherapy in Non-small Cell Lung Cancer
Brief Title: An Exploratory Study of Herombopag for Thrombocytopenia Induced by Chemotherapy Combined With Immunotherapy in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQBP-NSCLC-II-001
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- herombopag olamine tablets (Experimental)
  Interventions: Drug: herombopag olamine tablets

INTERVENTIONS:
Drug: herombopag olamine tablets — The first day of chemotherapy was d1, and the drug was started from d-5, 5 days before chemotherapy, with oral herombopag 5 mg/day for a maximum of 14 days. After chemotherapy, when the thrombocytopenia rises to ≥200×109/L, drug discontinuation can be considered

SUMMARY:
The purpose of this study is to explore the safety and efficacy of herombopag olamine tablets for thrombocytopenia induced by chemotherapy combined with immunotherapy in non-small cell lung cancer

DETAILED DESCRIPTION:
To observe and evaluate the safety and efficacy of the TPO receptor agonist herombopag for the secondary prevention of thrombocytopenia caused by chemotherapy combined with immunotherapy in non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the informed consent and voluntarily joined the study;
2. Age 18-75 years old, male or female;
3. Patients with stage IIIb-IV non-small cell lung cancer diagnosed by histopathology or cytology, who have received and will continue to receive carboplatin-based chemotherapy combined with pemetrexed or nab-paclitaxel, combined with immune checkpoint inhibitors ( ICIs) treatment;
4. The investigator determined that the patient could receive hetrombopag administration;
5. Thrombocytopenia of grade 2 or above occurred in the last chemotherapy cycle, defined as platelet count (PLT) ≤ 75×109/L;
6. The values of laboratory tests performed for screening shall meet the following criteria:

1) Blood routine examination: a) Hemoglobin (HB) ≥ 90 g/L; b) Absolute neutrophil count (ANC) ≥ 1.5×109/L; c) Platelet count (PLT) ≥ 80×109/L; 2) Biochemical tests: a) AST and ALT ≤ 3 times ULN (if there is tumor liver metastasis, ≤ 5 times ULN); b) TBiL ≤ 2 times ULN; c) Cr ≤ 2 times ULN, or creatinine clearance (CrCL) ≥60 mL/min (Cockcroft-Gault formula); 7. Life expectancy at screening ≥12 weeks; 8. ECOG: 0-1; 9. The main organ functions are normal, and there are no serious complications;

Exclusion Criteria:

1. pregnant or breastfeeding women;
2. Inability to understand the research nature of the research or to obtain informed consent;
3. The investigator judges other circumstances that are not suitable for inclusion in the study;
4. Thrombocytopenia caused by other causes other than those caused by chemotherapy or immunotherapy (such as chronic liver disease, sepsis, disseminated intravascular coagulation, immune thrombocytopenia, etc.);
5. Have unstable angina pectoris, congestive heart failure, uncontrolled hypertension, uncontrolled arrhythmia or recent (within 1 year of screening) history of myocardial infarction;
6. Those with a history of blood disease or tumor bone marrow infiltration;
7. Those who received concurrent radiotherapy and those who received pelvic radiotherapy in the past;
8. Arterial or venous thrombotic events within the past 6 months;
9. There are currently uncontrollable infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the response rate of hetrombopag | Follow-up to 28 days after the last use of herombopag
  response if all of the following criteria are met: 1. No need for platelet transfusion 2. No need to reduce chemotherapy drug dose due to thrombocytopenia 3. No need to delay chemotherapy due to thrombocytopenia) Note: chemotherapy drug dose reduction It was defined as reducing the dose of the original chemotherapy drug by ≥20%, and chemotherapy delay was defined as delaying chemotherapy by >7 days.

SECONDARY OUTCOMES:
The lowest platelet value after chemotherapy | Follow-up to 28 days after the last use of herombopag
  The lowest platelet value after chemotherapy
Platelet recovery to the highest value after chemotherapy; | Follow-up to 28 days after the last use of herombopag
  Platelet recovery to the highest value after chemotherapy;
The duration of platelets ≤50×109/L; | Follow-up to 28 days after the last use of herombopag
  The duration of platelets ≤50×109/L;
The time for platelets to recover to more than 100×109/L; | Follow-up to 28 days after the last use of herombopag
  The time for platelets to recover to more than 100×109/L;
Incidence of adverse events | Follow-up to 28 days after the last use of herombopag
  Incidence of adverse events

OTHER OUTCOMES:
Changes of platelet value in each visit cycle | Follow-up to 28 days after the last use of herombopag
  Changes of platelet value in each visit cycle

IPD SHARING:
Plan to Share IPD: No